CLINICAL TRIAL: NCT06412497
Title: MT2023-20: Hematopoietic Cell Transplant With Reduced Intensity Conditioning and Post-transplant Cyclophosphamide for Severe Aplastic Anemia and Other Forms of Acquired Bone Marrow Failure.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023LS101
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Severe Aplastic Anemia; Acquired Amegakaryocytic Thrombocytopenia; Acquired Pure Red Cell Aplasia; Paroxysmal Nocturnal Hemoglobinuria
Keywords: HCT; RIC; SAA; PTCy; aAT; aPRCA
MeSH Terms: conditions — Anemia, Aplastic; Acquired amegakaryocytic thrombocytopenia; Hemoglobinuria, Paroxysmal | interventions — Rituximab; thymoglobulin; Cyclophosphamide; fludarabine; Whole-Body Irradiation; Insulin Infusion Systems; Filgrastim; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: No clonal hematopoiesis (Experimental): Participants 25 years of age and younger with no clonal hematopoiesis. Active study treatment includes the conditioning regimen followed by the stem cell infusion and GvHD prophylaxis through day +180. Supportive care and follow up activities continue through two years post HCT.
  Interventions: Drug: Rituximab; Drug: Rabbit ATG; Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Biological: Cell Infusion; Drug: Post-Transplant G-CSF; Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- Arm B: Clonal hematopoiesis (Experimental): Participants 25-75 years old and/or with clonal hematopoiesis. Active study treatment includes the conditioning regimen followed by the stem cell infusion and GvHD prophylaxis through day +180. Supportive care and follow up activities continue through two years post HCT.
  Interventions: Drug: Rituximab; Drug: Rabbit ATG; Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Biological: Cell Infusion; Drug: Post-Transplant G-CSF; Drug: Tacrolimus; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Rituximab — For patients with EBV IgG seropositivity or EBV PCR positivity on pre-transplant evaluations, Rituximab 375 mg/m2 is given IV once on day -14 (+/-2 day) in the outpatient setting. Pre-medicate 30 minutes prior to rituximab with methylprednisolone (1 mg/kg) IV, acetaminophen 15 mg/kg (maximum 650mg) IV or PO and diphenhydramine 1 mg/kg (maximum 50mg) IV or PO.
Drug: Rabbit ATG — Rabbit ATG will be administered at doses and days indicated above, infused through a 0.22 micrometer filter over 4-6 hours. Pre-medicate 30 minutes prior to ATG infusion with methylprednisolone 1 mg/kg IV, (max dose = 125 mg), acetaminophen 15 mg/kg dose (max dose = 650 mg) enterally and diphenhydramine 1 mg/kg/dose (max dose = 50 mg) enterally or IV.
  Other Names: Thymoglobulin
Drug: Cyclophosphamide — Cyclophosphamide 14.5 mg/kg is be given as a 2-hour infusion on day -6. If the patient is obese (actual body weight (ABW) >/= 125% of the ideal body weight (IBW)), cyclophosphamide should be dosed using the adjusted body weight (AdjBW): 0.5(ABW-IBW) + IBW. Uroprotection with MESNA (14.5 mg/kg/day) in IV continuous infusion will be provided per institutional guidelines. Hyperhydration is not required for 14.5 mg/kg cyclophosphamide doses.
  Cyclophosphamide will be administered at 50 mg/kg using ABW over 2 hours on days +3 and +4. If the patient is obese (ABW >/= 125% of the ideal body weight (IBW)), cyclophosphamide should be dosed using the adjusted body weight (AdjBW): 0.5(ABW-IBW) + IBW. Uroprotection with MESNA (50 mg/kg/day) in IV continuous infusion as well as hyperhydration will be provided per institutional guidelines.
Drug: Fludarabine — For all patients, fludarabine dosing will be model-based using Bayesian methodology IV every 24 hours on days -6 to -3 with a cumulative area under the curve (cAUC) of 20 mg*hr/L.
Radiation: Total Body Irradiation — For patients age >/= 25 years, with myelodysplasia, or clonal hematopoiesis, total body irradiation will be 4 Gy, provided in two fractions on day -1. For all other patients, total body irradiation will be 2 Gy provided in a single fraction on day -1.
  Each dose of 2 Gy will be given at a dose rate between 1 and 1.9 Gy/minute prescribed to the midplane of the patient at the level of the umbilicus.
  Other Names: TBI
Biological: Cell Infusion — On day 0 the cells will be infused per cell source specific institutional guidelines.
Drug: Post-Transplant G-CSF — Beginning on day +5, patients will receive G-CSF SQ or IV 5 micrograms/kg once daily until post-nadir ANC > 1500/μL for 3 consecutive days or >3000/μL for 1 day.
  Other Names: Filgrastim
Drug: Tacrolimus — Tacrolimus will begin on day +5 at an initial dose of 0.03 mg/kg/day IV via continuous infusion. Goal trough levels will be 10-15 ug/mL until day +14 posttransplant, then decreased to a goal of 5-10 ng/mL thereafter. In the absence of GvHD, tacrolimus will discontinue at day +180 without a taper.
Drug: Mycophenolate Mofetil — Mycophenolate mofetil (MMF) therapy will begin on day +5. For pediatric service patients dosing of MMF will be 15 mg/kg/dose (max = 1000 mg) three times daily. For adult service patients dosing of MMF will be 15 mg/kg/dose (max = 1500 mg) twice daily. The same dosage is used orally or intravenously. Consider dose modification and/or pharmacokinetic measurements if renal and/or hepatic impairment (GFR<25 mL/minute corrected). Stop MMF at Day +35 or 7 days after engraftment achieved (ANC>500 x 106 neutrophils/L x 3 days) if later than day +35. If sufficient acute GvHD is observed to require systemic therapy, MMF should be continued for 7 days after initiation of systemic therapy. Afterward, use of MMF is at the discretion of the treating physician.
  Other Names: MMF

SUMMARY:
A phase II trial of a reduced intensity conditioned (RIC) allogeneic hematopoietic cell transplant (HCT) with post-transplant cyclophosphamide (PTCy) for idiopathic severe aplastic anemia (SAA), paroxysmal nocturnal hemoglobinuria (PNH), acquired pure red cell aplasia (aPRCA), or acquired amegakaryocytic thrombocytopenia (aAT) utilizing population pharmacokinetic (popPK)-guided individual dosing of pre-transplant conditioning and differential dosing of low dose total body irradiation based on age, presence of myelodysplasia and/or clonal hematopoiesis.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Severe Aplastic Anemia (SAA), characterized by one of the following:

  1. Refractory cytopenia(s), with 1+ of the following:

     1. Platelets <20,000/uL or transfusion dependent
     2. Absolute neutrophil count <500/uL without hematopoietic growth factor support
     3. Absolute reticulocyte count <60,000/uL AND bone marrow cellularity <50% (with < 30% residual hematopoietic cells)
  2. Early myelodysplastic features (bone marrow (BM) blasts <5%), without history of MDS/AML pre-treatment.
  3. Idiopathic SAA with post-HCT graft failure (blood/marrow donor chimerism <5%) requiring a 2nd allogeneic HCT
* Paroxysmal Nocturnal Hemoglobinuria (PNH), including AA-PNH overlap syndrome, acquired pure red cell aplasia (aPRCA), or acquired amegakaryocytic thrombocytopenia (aAT), characterized by one of the following:

  1. Refractory cytopenia(s), with 1+ of the following:

     1. Platelets <20,000/uL or transfusion dependent
     2. Absolute neutrophil count <500/uL without hematopoietic growth factor support
     3. Absolute reticulocyte count <60,000/uL or red cell transfusion dependent AND Bone marrow evidence of 1 to 3-lineage aplasia OR peripheral blood PNH clone >/= 10%
  2. Early myelodysplastic features (bone marrow (BM) blasts <5%) without history of MDS/AML pre-treatment.
  3. Idiopathic PNH, aPRCA, or aAT with post-HCT graft failure (blood/marrow donor chimerism <5%) requiring a 2nd allogeneic HCT
* Adequate organ function within 30 days of conditioning regimen

Exclusion Criteria:

* Pregnant, breastfeeding or intending to become pregnant during the study. Persons of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days of the start of treatment
* Uncontrolled infection
* Evidence of moderate or severe portal fibrosis or cirrhosis on biopsy
* Known allergy to any of the study components
* Prior radiation therapy deemed excessive by radiation therapist for proposed low dose TBI exposure on this protocol
* Diagnosis of an inherited bone marrow failure disorder such as Fanconi anemia, Telomere biology disorder, or Schwachman-Diamond syndrome, unless reviewed by the principal investigator and deemed appropriate for this approach (e.g. GATA2 deficiency)
* Advanced myelodysplastic syndrome (MDS; BM blasts >5%) or acute myeloid leukemia
* Psychiatric illness/social situations that, in the judgement of the enrolling Investigator, would limit compliance with study requirements
* Other illness or a medical issue that, in the judgement of the enrolling Investigator, would exclude the patient from participating in this study

Ages: 0 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2035-05-01 (Estimated); Study Completion 2036-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3-4 acute GvHD | 1 year post HCT
  Incidence of grade 3-4 acute graft-versus host disease (GvHD) at 1 year post HCT.
Incidence of chronic GvHD-free, failure-free survival (GFFS) | 1 year post HCT
  Incidence of chronic GvHD-free, failure-free survival (GFFS) 1 year post HCT
Incidence of chronic GvHD-free survival | 1 year post HCT
  Incidence of chronic GvHD-free survival at 1 year post HCT

SECONDARY OUTCOMES:
Incidence of failure-free survival (GFFS) | 2 years post HCT
  Incidence of chronic GvHD-free, failure-free survival (GFFS) 2 years post HC
Incidence of neutrophil recovery | Day 42 post HCT
  Incidence of neutrophil recovery at day 42 post HCT
Incidence of platelet recovery | 6 months post HCT
  Incidence of platelet recovery at 6 months post HCT
Incidence of grade 3-4 acute GvHD | 100 days post HCT
  Incidence of grade 3-4 acute GvHD at 100 days post HCT
Incidence of any chronic GvHD | 1 year post HCT
  Incidence of any chronic GvHD at 1 year post HCT
Overall survival | 1 and 2 years post HCT
  Overall survival at 1 and 2 years
Incidence of chronic GvHD-free survival | 2 years post HCT
  Incidence of chronic GvHD-free survival at 2 years post HCT

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States